CLINICAL TRIAL: NCT06251336
Title: Oral Supplementation With Uroial Plus in the Management of Infections and Urinary Symptoms Associated With Ureteral Stents.
Brief Title: Uroial Plus in the Management of Infections and Urinary Symptoms Associated With Ureteral Stents
Acronym: USSIAL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Foschi Nazario, Doctor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 6184
Record Dates: First submitted 2024-01-13; First posted 2024-02-09 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Ureteral Stent-Related Symptom; Urinary Tract Infections
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Intervention Model Description: 1:1
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Uroial Plus Arm (Experimental): UroialTM Plus sachets one sachet daily at night before going to bed after urinating for 30 days
  Interventions: Other: UroialTM Plus
- Placebo Arm (Placebo Comparator): one placebo sachet daily at night before going to bed after urinating for 30 days
  Interventions: Other: Placebo

INTERVENTIONS:
Other: UroialTM Plus — Nutraceutical
  Other Names: UroialTM Plus S&R Pharmaceutics S.p.A.
  Arms: Uroial Plus Arm
Other: Placebo — Placebo sachet
  Arms: Placebo Arm

SUMMARY:
Double-blind randomised interventional pilot study. To evaluate whether therapy with UroialTM Plus has a role in rebalancing homeostasis in ureteral stent patients, improving symptoms related to the presence of the ureteral stent in place.

Ureteral stent patients will be randomised into two groups:

* the experimental group will receive UroialTM Plus sachets, one sachet daily at bedtime after urinating, for 30 days
* the control group will receive a placebo, one sachet daily in the evening before going to bed after urinating, for 30 days.

At each visit, the investigator will assess the possible occurrence of urinary symptoms, their severity and their impact on quality of life by administering the following questionnaires: IPSS, USSQ, AIA, SF-36, VAS, EQ-5D-5L.

DETAILED DESCRIPTION:
Study design The study is a pilot, interventional, double-blind, randomised clinical trial for two parallel groups with an intervention allocation ratio of 1:1. In this way it will be possible to evaluate the role of UroialTM Plus in rebalancing homeostasis in patients with ureteral stents, compared to a group of subjects, also with ureteral stents, who will be given a placebo. Data will be collected by filling in specific questionnaires by patients. The evaluation of the results of the questionnaires will be carried out in blind by an external operator.

Duration The study will last 16 months including a 12-month enrolment period. The study will start after the ethics committee has given a favourable opinion.

Setting The study will be conducted at the U.O.C of the Urological Clinic of the Policlinic "A. Gemelli" in Rome.

METHODS Population Seventy-eight patients undergoing ureteral stent placement after endourological treatment for calculosis or abdominal surgery will be consecutively enrolled at the Urology Clinic of the same hospital.

Patients will be assessed at the time of recruitment and subsequently re-evaluated at 7 and 30 days after enrolment.

INTERVENTIONS Patients eligible for enrolment will be assessed by specialists in endourology and the treatment of urinary stones. The severity of lower urinary tract symptoms will be assessed using the International Prostatic Symptoms Score (IPSS) and the Ureteral Stent Symptom Questionnaire (USSQL). Concurrently, the investigator will assess the impact on quality of life and impairment of daily activities using the Activity Impairment Assessment (AIA), the Short Form 36 Questionnaire (SF- 36), the Visual Analogue Scale (VAS) and the EuroQol Group Questionnaire (EQ-5D-5L).

Ureteral stent patients will be randomised into two groups:

* the experimental group will receive UroialTM Plus sachets, 1 sachet daily at night before going to bed after urinating, for 30 days
* the control group will receive a placebo, 1 sachet daily in the evening before going to bed after urinating, for 30 days At each visit, the investigator will assess the possible occurrence of urinary symptoms, their severity and their impact on quality of life by administering the following questionnaires: IPSS, USSQ, AIA, SF-36, VAS, EQ-5D-5L.

Demographic characteristics of all enrolled patients will also be collected. Patients will subsequently be re-evaluated at 7 and 30 days after enrolment.

RANDOMISATION A permuted block randomisation of subjects will be performed by an operator using online software to provide the permuted random blocks. Symptom assessment questionnaires self-administered to patients at follow-up visits will be kept in sealed and sequentially numbered opaque envelopes, which will be guarded by the same operator and will not contain any patient master data. Both operators and patients will not be aware of the allocation to the groups, and an external investigator will carry out the evaluation of the self-administered questionnaires to the patients, without being aware of which patient belongs to the treatment group and which to the control group.

INSTRUMENTS The IPSS is a questionnaire aimed at objectively assessing the urinary symptoms of patients with prostatic hypertrophy. It consists of 8 questions with 6 possible answers indicating increasing severity of the symptom. The score ranges from 0 to 35 (from symptomatic to very symptomatic). Higher scores indicate more severe symptoms. Scores below seven are considered mild.

The USSC is a questionnaire used to assess the influence of the presence of ureteral stents on several health domains concerning urinary symptoms, pain, general health, impact on work activities, sexuality and other daily problems. It consists of 6 sections and 38 items.

The AIA scale will be used for the assessment of impairment of daily activities related to urinary symptoms during infection. It consists of 5 items with 5 possible responses per item (0-4), the higher the score the greater the impairment of daily activities.Short Form 36 (SF-36) is a questionnaire that aims to quantify health status and measure health-related quality of life, allowing the impact of a disease on various dimensions of quality of life to be captured. It consists of 36 questions that can be divided into 8 scales. All items have the same response mode using a scale with a variable weighted score for each item. Each of the 8 summed scores is transformed linearly on a scale from 0 (negative health) to 100 (positive health).

Pain intensity will be assessed using the Visual Analogue Scale (VAS), which corresponds to a predetermined line 10 cm long, where the left end corresponds to 'no pain' and the right end to 'worst possible pain'. The patient will be asked to draw a mark on the line representing the level of pain experienced.

EuroQol Group Questionnaire (EQ-5D-5L) assesses health status by means of severity scales for five aspects (mobility, personal care, performance of daily activities pain/discomfort, anxiety/depression). Each dimension has three levels of response (no problems, some problems, many problems) The data will be reported on a dataset by the external investigator. SAMPLE SIZE The sample size is calculated on the basis of scientific evidence reporting the presence of ureteral stent-related symptomatology in more than 80% of patients with ureteral stents.

With an estimated standardised effect size of 0.57, an alpha error of 5% and a main trial power of 80%, 39 patients per group are required for a total of 78 patients.

STATISTICAL ANALYSIS Patient demographic, clinical and laboratory variables will be summarised using descriptive statistical techniques. In particular, quantitative variables distributed as a normal will be reported as mean and standard deviation (SD) otherwise as median and interquantile range (IQR). Qualitative variables will be reported as absolute and relative (percentage) frequencies. Analyses will be performed overall and stratified by treatment groups.

The assumption of normality of the quantitative variables will be checked by means of the Shapiro- Wilks test.

Categorical variables will be compared by means of the Chi-square test and/or Fisher's exact testThe difference in mean of the quantitative variables measured at two time instants, within each group, will be tested by applying Student's t-test for paired data or Wilcoxon's test.

Keeping time fixed, the comparison between the two groups for all analysed parameters will be performed by employing Student's t-test and/or the Mann-Whitney test.

A mixed-effects model for longitudinal data (GLMM) will be fitted to evaluate changes in the variables of interest over time taking the group effect into account. In addition, potential confounding factors will be included in the model.

Results will be considered statistically significant when p-values < 0.05. All analyses will be performed using the statistical programme STATA (version 14).

SAFETY / ADVERSE EVENT MANAGEMENT All adverse events observed during the study will be collected and recorded. Suspected adverse reactions from dietary supplements will be reported through the online phytovigilance system ''VigiErbe'' managed by the Institute of Sanity, in collaboration with AIFA and the Ministry of Health

SAFETY REFERENCE DOCUMENT Descriptive sheet of the products under study.

ETHICAL CONSIDERATIONS The study will be conducted in accordance with Good Clinical Practice. All patients will provide written informed consent. The study protocol will be evaluated by the Ethics Committee Territorial.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* patients with ureteral stents after endourological treatment for stone disease or abdominal surgery
* ability to sign informed consent

Exclusion Criteria:

* positive urine culture 1 month before enrolment
* recurrent urinary tract infections (3 episodes in the last 12 months, or 2 episodes in the last 6 months)
* previous pelvic radiotherapy
* history of transitional cell carcinoma (TCC)
* history of painful bladder syndrome, actinic cystitis, chronic pelvic pain
* symptomatic benign prostatic hypertrophy under treatment (for males)
* presence of indwelling bladder catheter, suprapubic cystostomy, percutaneous nephrostomy, percutaneous cystostomy, urinary diversion
* pregnancy or lactation
* life expectancy < 1 year
* patients unable to give or refusing to sign informed consent
* inability to follow protocol procedures
* any condition that the investigator believes may be hazardous to the health of the Patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Improvement rate | 30 days after recruitment
  Improvement rate will be the main endpoint of the study, and is defined as improvement of symptoms related to the presence of the ureteral stent with evidence to the answers of the questionnaires

SECONDARY OUTCOMES:
Recruitment feasibility | 30 days after recruitment
  Percentage of patients who complete the study. It will measured by counting empty Uroial TM Plus sachets at the scheduled visit
Complications | 30 days after recruitment
  The number of admissions to the emergency room for symptoms not responsive to standard therapy.
Impact on employment | 30 days after recruitment
  The number of working days lost for symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Nazario Foschi, MD, Principal Investigator — Università Cattolica del Sacro Cuore, Policlinico Universitario Agostino Gemelli

IPD SHARING:
Plan to Share IPD: No